CLINICAL TRIAL: NCT04617106
Title: Palpation Versus Ultrasound-guided Dynamic Needle Tip Positioning Technique for Radial Artery Cannulation in Adult Surgical Patients
Brief Title: Radial Artery Cannulation Using Two Different Methods.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Dr Sujan Dhakal, Resident Doctor, PGY II, Anesthesia and Critical care, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 686-2020
Record Dates: First submitted 2020-10-22; First posted 2020-11-05 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Radial Artery Cannulation

STUDY DESIGN:
Intervention Model Description: In patients undergoing elective surgery who need arterial catheter placement, radial artery cannulation will be done using either the conventional palpation method or USG-guided dynamic needle tip positioning method before the induction of anaesthesia. In one group, radial artery cannulation will be done using the conventional palpation method, and in the second group, USG-guided dynamic needle tip positioning method will be employed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Palpation group (Active Comparator): In patients undergoing elective surgery who need arterial catheter placement, radial artery cannulation will be done using the conventional palpation method.
  Interventions: Procedure: Radial artery cannulation
- DNTP group (Active Comparator): In patients undergoing elective surgery who need arterial catheter placement, radial artery cannulation will be done using USG-guided dynamic needle tip positioning method.
  Interventions: Procedure: Radial artery cannulation

INTERVENTIONS:
Procedure: Radial artery cannulation — cannulation of Radial artery using standard IV cannula (axillary drug port will be taped using opaque adhesive)

SUMMARY:
Radial Artery cannulation using conventional palpation vs USG guided Dynamic needle tip positioning (DNTP) method.

DETAILED DESCRIPTION:
Management protocol of patients

A day before surgery All the patients included in the study will be explained in detail about the purpose of the study, and the need, benefits, and risks of arterial cannulation and the purpose of the study.

Written informed consent will be obtained during the pre-anaesthetic checkup. Patients will be asked to remain nil per oral as per standard American Society of Anesthesiologists guidelines. Premedication will be advised as per institutional protocol.

Pre-anaesthetic room After shifting from the ward to the pre-anaesthetic room, an intravenous line will be secured with an 18 or 20 G cannula in the dominant hand and baseline heart rate, blood pressure and oxygen saturation will be recorded. The patient will then be shifted to the operation theatre.

Operation theatre After shifting to the operating table, a pulse oximeter, a non-invasive blood pressure monitor, and an electrocardiogram monitor will be attached.

Arterial pressure transducer and tubings will be flushed with normal saline and will be kept ready.

Barbeaue test will be done using pulse oximetry in the thumb of the non-dominant hand to assess the type of Ulnopalmar arch.

The anaesthesia faculty/resident/assistant not involved in the study will then be asked to open an opaque, sealed envelope to decide the technique to be used for cannulation.

Radial artery cannulation Radial artery catheterisation will be done by the investigating anaesthesiology resident under the supervision of the consultant anaesthesiologist in the operation theatres.

The anaesthesia resident performing arterial cannulation must have placed at least 20 radial arterial catheters by palpation method and 20 using USG-guided DNTP method.

The patient's arm will be slightly abducted (less than 90 degrees) from the body and placed on an arm board and the wrist will be placed in an extended position by placing a towel roll making an approximately 60-degrees angle with the forearm. The wrist will be then stabilised in this position by taping it to the arm board.

To maintain asepsis, the wrist will be then prepped with povidone Iodine 10%. Surgical gloves, sterile drapes, and a sterile plastic sheath for USG-guided technique will be used.

The investigating resident will sit on a chair of a comfortable height facing the patient's wrist.

To anaesthetise the cannulation site, 1 ml of 2% lidocaine will be injected with a 25-gauge needle, approximately 3 cm proximal to the distal wrist crease after wiping off the povidone iodine with a sterile gauge.

A 20-Gauge intravenous catheter of the same trademark will be used to catheterise the radial artery in all patients.

The timer (SEIKOSHA stopwatch, Seikosha co. ltd, Japan) will be started once the USG-probe is placed on the prepped wrist or when the operator begins palpation of the radial pulse in the USG-guided and palpation techniques, respectively.

Immediately after successful cannulation, an assistant will attach the pressure monitoring tubing.

The timer will be immediately stopped once the arterial waveform appears on the monitor.

If after 300 seconds, the radial artery is not cannulated, the procedure will be aborted, and documented as "failure to cannulate." A senior anaesthesiologist will then perform arterial cannulation using any method at his/her discretion.

Following data will be collected Systolic and diastolic blood pressure before cannulation using NIBP First pass success of radial cannula placement Number of cannulae used Number of skin punctures Number of redirections Time for successful cannulation (in secs)

USG guided DNTP technique USG machine (Sonosite M-Turbo, Fujifilm Sonosite Inc. USA) with a linear probe (6-13 MHz) will be used, using the vascular mode, optimal gain, and autofocus.

A short-axis out-of-plane view of the radial artery will be obtained and kept at 1.5 cm depth aligned with the central line of the USG probe.

The needle and catheter will be advanced through the skin at an angle of 45 to 60 degrees until the hyperechoic needle tip is seen on the ultrasound image.

The ultrasound probe will then be moved proximally along the forearm and away from the needle insertion point until the needle tip disappears from the ultrasound image.

The needle and catheter will then be advanced a few millimeters until the needle tip is seen again on the ultrasound image.

This stepwise process will be repeated several times until the needle tip is visualised in the lumen of the radial artery.

At this point, the angle of approach will be decreased and the same process shall be continued, keeping the needle tip in the center of the arterial lumen.

The needle and catheter assembly will be advanced stepwise for approximately 3 to 5mm inside the arterial lumen.

If the needle is advanced through the posterior vessel wall, the operator will be allowed to withdraw the needle slightly and advance again.

After around 3 to 5mm of the needle is advanced, the catheter will then be threaded off the needle and the pressure-monitoring tubing will be immediately attached.

Palpation method The investigating resident will palpate the radial arterial pulse with the non-dominant hand.

The needle and catheter assembly will be advanced towards the radial artery at a 15° to 30° angle until a flashback of blood is observed in the needle hub.

Once flash-back of blood appears in the hub, the needle angle will be decreased slightly and the catheter will be advanced about 3 to 5mm.

If the operator suspects puncture of the posterior arterial wall, the cannula will then be gradually withdrawn such that the cannula tip will be in the arterial lumen. The intraluminal position of the catheter will be ensured by blood in the catheter lumen as the needle is being withdrawn. The needle angle will then be decreased slightly and the catheter will be advanced.

If blood continues to flow into the hub, the catheter will be threaded off the needle and then the pressure-monitoring tubing will be attached.

A new cannula will be used if the cannula hub is full of blood but the artery is not cannulated successfully or there is obvious catheter kinking or shearing during redirections or skin punctures.

After radial artery cannulation Once radial artery cannulation is complete, the cannula will be secured with adhesive tape and injection port will be covered with an opaque dressing to prevent inadvertent intra-arterial injection of drugs.

The wrist will then be placed in a neutral position with the forearm placed either parallel to the torso or abducted and secured on an arm board.

Routine preoxygenation, anaesthesia induction, patient positioning, and maintenance of anaesthesia will be done as per standard institutional practice.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective surgeries Patients who require arterial cannulation as determined by the consultant anaesthesiologist Age: 18 years or above

Exclusion Criteria:

Type D ulnopalmar arch patency during Barbeau test Patient with a documented history of peripheral vascular disease Infection or other soft tissue lesions at the site of cannulation A surgical procedure involving the cannulation site Patients receiving inotropes or vasopressors.

* History of radial artery cannulation within the past one month at the planned cannulation site.
* Patients with an arterial catheter in-situ (any site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
First pass success rate between conventional palpation method with USG-guided DNTP method | through study completion, an average of 6 months
  compare the successfully obtaining an arterial waveform with a single skin puncture, irrespective of the number of needle re-directions needed.

SECONDARY OUTCOMES:
To compare the number of skin punctures between conventional palpation method with USG-guided DNTP method | through study completion, an average of 6 months
  puncture in the skin made by the cannula in an attempt to cannulate the radial artery will be assessed between the groups
To compare the number of cannulae used for successful radial artery cannulation between conventional palpation method with USG-guided DNTP method | through study completion, an average of 6 months
  number of cannula required for successful cannulation between two groups will be compared
To compare the time duration for successful cannulation in conventional palpation method with USG-guided DNTP method | through study completion, an average of 6 months
  total time (in seconds) taken from the placement of USG-probe on the prepped wrist or when the operator begins palpation of the radial pulse to the appearance of the arterial waveform in the monitor will be compared between two groups
To compare overall five-minute success rate in conventional palpation method with USG-guided DNTP method. | through study completion, an average of 6 months
  overall success between two groups after 5 minutes will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuwan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: data will be available within 2 months of completion of study, around August 2021. It will be available for 2yrs form the time of completion of study.
Access Criteria: anyone interested in similar research can access.